CLINICAL TRIAL: NCT00540735
Title: Efficiency Evaluation of Photodynamic Therapy With Photofrin® on Unresectable Type III or IV Cholangiocarcinomas - A Prospective, Multicentric and Randomized Study.
Brief Title: Efficiency Evaluation of Photodynamic Therapy With Photofrin® on Unresectable Type III or IV Cholangiocarcinomas
Acronym: CK/PDT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Big difficulties to enroll patients
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 2006-01
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2007-10

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): PDT
  Interventions: Procedure: photodynamic therapy
- 2 (No Intervention)

INTERVENTIONS:
Procedure: photodynamic therapy
  Arms: 1

SUMMARY:
Unresectable type III or IV cholangiocarcinoma has a very bad prognosis; survival median ranges between 6 and 9 months.

Survival depends on biliary drainage quality, obtained by plastic or metallic prothesis setting up in one or several hepatic segments.

Radiotherapy and/or chemotherapy didn't prove yet their efficiency on survival. In France, gemcitabin is recommended by the French Digestive Oncology Federation in metastatic tumours, in monotherapy or associated with cisplatin or oxaliplatin (Gemox) for patients in good general condition.

Photodynamic therapy has shown in 3 prospective studies - one randomized - with small patient series, a significative efficiency on survival and quality of life of treated patients, in comparison with historical series, or patients' groups whose biliary drainage was in most cases unefficient.

A new randomized study, including patients whose biliary drainage is efficient and comparing their becoming when they are treated by PDT in addition to current practice, or only by current practice, seems to be justified.

The principal objective of this study is to evaluate the efficiency of PDT with Photofrin® on patients with unresectable type III or IV cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Obtention of a written informed consent.
* Patient over 18.
* Patient with a type III or IV (according to Bismuth classification) histologically proved cholangiocarcinoma ; histologic diagnosis must be proved by biliary brushing, bile cytology, endobiliary biopsy under scope control with pediatric pliers, or by cytologic puncture under scan or echoendscopic control.
* Patient with Karnofsky score ≥ 50 %
* Patient with an efficient initial biliary drainage with prothesis.
* Cancer classified maximum T3N1M1, but only with intrahepatic metastasis occupying less than 25% of hepatic parenchyme (according to TNM cancer classification of extrahepatic biliary ducts' cancers).
* Patient capable of fill in the quality of life questionnaire.

Exclusion Criteria:

* No written informed consent.
* Type I and II cholangiocarcinoma according to Bismuth classification.
* Patients with ASA score 4.
* Patients with clinical and biological signs of biliary infection.
* Patients with a severe visceral disease other than cholangiocarcinoma.
* Patients without an efficient initial biliary drainage.
* Patients with extrahepatic visceral metastasis, except perihilar ganglionic metastasis classified T4N1M+ according to TNM classification.
* Patients whose cholangiocarcinoma has already been resected.
* Patients under or already treated by radiotherapy or chemotherapy treatment for cholangiocarcinoma.
* Patients first treated with metallic prothesis.
* Patients with a contraindication to MRI.
* Patients with porphyria or hypersensibility to porphyrins.
* Patient treated by a non authorized treatment at the time of inclusion.
* Pregnant, parturient or breastfeeding women.
* Non menopaused woman without an efficient contraception.
* Patient under 18.
* Person over 18 under protection according to French Public Health Code.
* Person not affiliated to a social security regimen, or benefiting from such a regimen.
* Person in a exclusion period of another biomedical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2008-04; Study Completion 2009-11

PRIMARY OUTCOMES:
Patients' survival compared between both groups : PDT and non-PDT.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Boyer, MD, PhD, Principal Investigator — UH Angers
Locations (18):
- France (18):
  - UH Amiens, Amiens
  - UH Angers, Angers
  - H Beaujon, Clichy
  - UH Henri Mondor, Créteil
  - UH Kremlin Bicêtre, Le Kremlin-Bicêtre
  - UH Claude Huriez, Lille
  - Clinique Sainte Anne, Lyon
  - UH La Timone, Marseille
  - UH Marseille Nord, Marseille
  - H Metz-Thionville, Metz
  - UH Nantes, Nantes
  - Clinique du Trocadéro, Paris
  - UH Cochin, Paris
  - UH La Milétrie, Poitiers
  - UH Charles Nicolle, Rouen
  - UH Hôpital Civil, Strasbourg
  - UH Purpan, Toulouse
  - UH Rangueil, Toulouse